CLINICAL TRIAL: NCT06175377
Title: Antiplatelet Therapy After Successful Percutaneous Coronary Intervention for Chronically Occluded Coronary Artery: A Prospective, Multicenter, Randomized Study Comparing Two Durations of Dual Antiplatelet Therapy
Brief Title: Antiplatelet Therapy After Successful Percutaneous Coronary Intervention for Chronically Occluded Coronary Artery
Acronym: DAPT-CTO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCAPHM23_0327
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Chronic Total Occlusion
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long dual Aspirin/Clopidogrel therapy (Active Comparator): Patients will be treated with usual long dual antiplatelet aggregation for 6 to 12 months
  Interventions: Procedure: Percutaneous coronary intervention; Other: Long dual Aspirin/Clopidogrel therapy; Other: Follow-up visit at 1 month; Other: Follow-up visit at 6 months; Other: Follow-up visit at 12 months
- Short dual Aspirin/Clopidogrel therapy (Experimental): Patients will be treated with short dual antiplatelet aggregation for 1month
  Interventions: Procedure: Percutaneous coronary intervention; Drug: Short dual Aspirin/Clopidogrel therapy; Other: Follow-up visit at 1 month

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — A percutaneous coronary intervention for chronic total occlusion lesion with at least one implanted coronary stent will be performed as part of routine care.
Drug: Short dual Aspirin/Clopidogrel therapy — Aspirin will be prescribed as part of the patient's normal course of care, according to current recommendations. The second antiplatelet agent will be clopidogrel, the duration of which will vary according to the randomization group of each patient included. Patients will be treated for 1 month.
  Arms: Short dual Aspirin/Clopidogrel therapy
Other: Long dual Aspirin/Clopidogrel therapy — Aspirin will be prescribed as part of the patient's normal course of care, according to current recommendations. The second antiplatelet agent will be clopidogrel, the duration of which will vary according to the randomization group of each patient included. Patients will be treated for 6 to 12 months.
  Arms: Long dual Aspirin/Clopidogrel therapy
Other: Follow-up visit at 1 month — At 1 month following the inclusion a visit or a phone call with the referring cardiologist will be organized.
Other: Follow-up visit at 6 months — At 6 months following the inclusion a visit or a phone call with the referring cardiologist will be organized.
  Arms: Long dual Aspirin/Clopidogrel therapy
Other: Follow-up visit at 12 months — At 12 months following the inclusion a visit or a phone call with the referring cardiologist will be organized.
  Arms: Long dual Aspirin/Clopidogrel therapy

SUMMARY:
Coronary arteries are in charge of oxygen supply for the myocardium. When coronary arteries develop stenosis the coronary blood flow (i.e. oxygen flow) is reduced. Chronic total occlusion (CTO) is the extreme evolution of a coronary stenosis, which ends up to a total vessel closure.

Percutaneous coronary intervention (PCI) is the main treatment for chronic occlusions. The principle of this treatment is to implant a stent covering the whole segment of occlusion and allowing the blood to perfuse the myocardium antegradely and not retrogradely via the collateral(s). This angioplasty and stent implantation requires a dual antiplatelet therapy (aspirin associated with clopidogrel) to prevent a new thrombosis within the newly placed coronary stent.

Following the development of coronary stent (and particularly drug eluting coronary stent) new thrombosis within the implanted coronary scaffold have emerged. Dual antiplatelet therapy (DAPT) (compared to single antiplatelet therapy or anticoagulant) and initially prolonged DAPT (12 months) has offered a preventive treatment for stent thrombosis after PCI.

PCI treatment for CTOs continues to increase in France and around the world, while no dedicated study has been proposed so far regarding DAPT duration. Therefore, the general European recommendations for DAPT in chronic coronary syndrome management guidelines should be applied even though the CTO poses specific technical challenges (long and multiple stenting length for example). Even if 6 months DAPT is recommended as routine duration in chronic coronary syndrome (CCS), longer DAPT (12 months) is possible in this setting. However, the optimal duration of DAPT is not clearly demonstrated on an individual basis and each physician must adapt the DAPT duration for each single patient. A so called "ischemic / bleeding balance "guides the duration of DAPT.

This study would be the first randomized protocol to clarify the efficacy and safety of a shorter DAPT duration in the specific context of CTO PCI. It is conceivable that the technical advances which have made it possible to reduce the duration of DAPT to up to 1 month, in the cases of patients at high risk of bleeding for example, could be applicable to CTO PCI. Therefore, reducing the DAPT to 1 month, in the setting of CTO PCI, could reduce the haemorrhagic risk which should be proportional to the duration of the DAPT. Moreover, the invesitgators will evaluate the safety of short DAPT in terms of ischemic events during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a successful coronary stent implantation for chronic coronary occlusion, eligible for long-term aspirin therapy and requiring a dual antiplatelet therapy
* Affiliated to Social Security system.
* Signature of informed consent.
* Age > 18 years old.

Exclusion Criteria:

* Dual antiplatelet therapy contra-indication
* Patient with hypersensitivity to aspirin (or any of its excipients) and/or to any of the active substance or to any of the excipients of the investigational medical product used in this study (clopidogrel);
* Patient with contraindication to aspirin and/or clopidogrel.
* No coronary stent implanted
* Age < 18years
* Patient under guardianship
* Pregnancy or breast feeding
* Prasugrel or ticagrelor use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
bleeding events at 12 months | 12 months
  time-to-composite endpoint of bleeding events will be assessed according to the Bleeding Academic Research Consortium (BARC) Classification (BARC2 to BARC5) during follow-up (12 months).
ischemic events at 12 months | 12 months
  time-to-composite endpoint of ischemic events (all cause death, stroke, stent thrombosis, myocardial infarction, repeat revascularization, rehospitalisation for angina) will be recorded during follow-up (12 months).

SECONDARY OUTCOMES:
Major adverse ischemic clinical events (MACE) | 12 months
  time-to-composite endpoint of ischemic stroke, cardiovascular death, stent thrombosis, repeat revascularization, rehospitalisation for angina over 12 months follow-up, taking into account the competing risk of death from non-cardiovascular cause, or time to last follow-up in case of no MACE
Time-to-bleeding | 12 months
  Time-to-bleeding event defined according to Bleeding Academic Research Consortium (BARC) classification (BARC 2 to BARC 5) over 12 months follow up, taking into account the competing risk of death from non-haemorrhagic cause, or time to last follow-up in case of no bleeding event.The BARC classification goes from 0 (no bleeding) to 5b (Fatal bleeding. Overt bleeding, autopsy, or imaging confirmation).
Time-to-all cause death | 12 months
  Time-to-all cause death over 12 months follow-up, or time to last follow-up in case of no death
Compliance to drug regimen at 1 month | 1 month
  Compliance to drug regimen at will be assessed by telephone or during an clinical visit 1 months after the inclusion
Compliance to drug regimen at 6 months | 6 months
  Compliance to drug regimen at will be assessed by telephone or during an clinical visit 6 months after the inclusion
Compliance to drug regimen at 12 months | 12 months
  Compliance to drug regimen at will be assessed by telephone or during an clinical visit 12 months after the inclusion

IPD SHARING:
Plan to Share IPD: No